CLINICAL TRIAL: NCT06486714
Title: Mechanical Alignment Versus Kinematic Alignment Total Knee Arthroplasty: A Randomized Control Trial
Brief Title: Mechanical Alignment Versus Kinematic Alignment Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 217306
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Our study will randomize patients to receive either cemented MA-TKA or KA-TKA with the goal of assessing pain scores and PROMs at various time points following surgery.
Who Masked: Participant
Masking Description: Single blind. The participant will be blinded to the assignment until one year after surgery. The study team and surgeon will not be blinded to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinematic Total Knee Arthroplasty (Experimental): KA-TKAs recreate the native joint line, hip-knee-ankle angle, and rotation of the pre-arthritic joint.
  Interventions: Procedure: Total knee arthroplasty
- Mechanical Total Knee Arthroplasty (Active Comparator): MA-TKAs are performed by which the distal femur and proximal tibia cuts are made perpendicular to the mechanical axis, a line connecting the center of the femoral head to the center of the ankle. These cuts are classically described as a 6-degree valgus cut of the distal femur and a 0-degree cut of the proximal tibia in relation to the mechanical axis. MA-TKAs create a 0-degree hip-knee-ankle angle.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — All patients indicated for primary total knee arthroplasty will receive a cruciate-retaining cemented or cementless implant system, utilizing either MA or KA methodology.

SUMMARY:
Historically, total knee arthroplasty (TKA) has been performed with the goal of restoring a neutral mechanical axis, eliminating the average 3 degrees of valgus and varus of the distal femur and proximal tibia joint lines respectively. This is thought to provide a more stable and neutral joint-bearing surface. Because of this shift to a 0-degree knee angle, soft tissue releases are frequently required to balance the knee after making the distal tibia and proximal tibia cuts. More recently and increasingly, TKAs have been performed with a goal of restoring kinematic, or anatomic, alignment of the knee. This is thought to provide a more normal native knee angle, with the hopes of precluding the necessity of soft tissue releases to balance the knee. While some studies are promising regarding kinematically aligned TKAs (KA-TKA), at present, it is unclear how these compare to mechanically aligned TKAs (MA-TKA) in terms of patient reported outcome measures (PROM) when compared head-to-head.

This study will randomize patients to receive either cemented MA-TKA or KA-TKA with the goal of assessing pain scores and PROMs at various time points following surgery.

DETAILED DESCRIPTION:
Participants include patients 18 years or older presenting to the the investigators' institutions indicated for a primary total knee arthroplasty. Exclusion criteria include revision TKA, patients with prior injuries to study knee, patients with history of childhood knee disease, patients who cannot complete questionnaires in English, patients with comorbidities preventing surgery, and patients who are not able to provide informed consent.

If, after examination, the patient is still eligible, the surgeon will introduce the study. If the patient is receptive, a member of the study team will approach the prospective patient to explain the study in detail. The study team members will emphasize the voluntary nature of participation and the prospective participant will be encouraged to ask questions and speak to others about participation. Once questions are answered to the prospective participant's satisfaction, they will be presented with the informed consent document (ICD). The study team member will exit the exam room to allow the prospective participant to carefully read the consent form. If they wish, prospective participants will be provided with a paper copy of the ICD to read and discuss with whomever they wish. Once the study team member and surgeon, if required, have answered any additional questions, the participant will sign the ICD. Preferably, the ICD will be signed in clinic. If a prospective participant has taken then ICD with them to consider or discuss with others, a study team member will plan a time to meet the prospective participant in the Orthopaedic Surgery clinic (likely in the preoperative holding area) to sign the ICD and complete the baseline questionnaires and ROM. Patients will have up until the day of surgery to decide if they would like to participate in the study.

Informed consent will be obtained from participants before surgery. Preferably, the ICD will be signed in clinic. If a prospective participant has taken then ICD with them to consider or discuss with others, a study team member will plan a time to meet the prospective participant in the Orthopaedic Surgery clinic (likely when they return for preoperative clearance) to sign the ICD and complete the baseline questionnaires and ROM. Shortly after the ICD is signed, the participant will be randomized to either receive MA-TKA or KA-TKA. The participant will be blinded to the assignment until one year after surgery. The study team and surgeon will not be blinded to the assignment. Randomization will occur using stratified randomization lists per site. The Biostatistics Core at the Loyola University Clinical Research Office will provide randomization lists for each site to ensure equal 1:1 allocation of the two methods within each institution. Loyola Biostatistics will ensure randomization lists are readily available via REDCap at the time of consent/randomization. A member of the study team will communicate the randomization assignment to the surgeon and/or surgery scheduler. Preoperative instruction, surgery, and postoperative care/instructions will be the same for study participants as for patients who are not participating in the study. Two weeks after surgery, participants will return to the clinic for standard of care postoperative examination. The participant will be asked to complete questionnaires using a Loyola-managed electronic device. If desired, the participant can also request that a link to the questionnaires be emailed ahead of their appointment to be completed on their own device. Participants will also be asked to complete the same questionnaires prior to or at their standard 6-week postoperative visit and at the standard of care 1-year postoperative visit.

All patients indicated for primary total knee arthroplasty will receive a cruciate-retaining cemented or cementless implant system, utilizing either MA or KA methodology. Both TKA types have been proven successful clinically and in the literature. A placebo would not be appropriate or ethical. Participants will be blinded to the assignment until one year after surgery. The study team and surgeon will not be blinded to the assignment.

The primary aim of the study will be measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function and Pain Interference item banks, the Knee Injury and Osteoarthritis Outcome Score (KOOS) Jr., the Forgotten Joint Score, and a validated 0-10 visual analog scale (VAS) of patient pain. KOOS Jr scores at 6 weeks post operation will be considered the primary endpoint. Secondary aims include evaluating KOOS Jr at 2 weeks and 1 year postoperatively. In addition to KOOS Jr, postoperative opioid consumption, pain scores, self-reported outcomes, range of motion, and survivorship will be collected at all time points.

A 10-point difference in KOOS score is deemed clinically relevant between KA-TKA and MA-TKA methods. Using previously published data, KOOS has a conservative standard deviation estimate of 18. Using an independent sample t-test with 80% power and a 2-sided alpha value of 0.05, a sample size of 48 independent patients per method is sufficient to test the null hypothesis of no difference in KOOS, with an alternative hypothesis of +/- 10 points difference. With possible attrition of 5%, this sample size is inflated to 51 per group.

The investigators' hypothesis is that patients with KA-TKAs will have higher PROMs compared to patients who receive MA-TKAs.

MA-TKAs and KA-TKAs are commonly used procedures. Both procedures will be performed in a standard of care manner. There is no additional surgery risk to participants when participating in this study. Subject safety will be monitored like any other patient receiving a total knee arthroplasty by post-operative visits, patient-reported outcome measures, radiographic studies, and access to a contact number should patients have questions/concerns. Patients may experience a loss of confidentiality because of study participation. The frequency of this risk is rare. We do not expect any increased failure rate in either group as many studies have shown both techniques to be safe and efficacious. However, if there is a dramatic difference in failure rate our outcomes, we will halt the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older presenting to our institutions indicated for a primary total knee arthroplasty

Exclusion Criteria:

* Revision TKA
* Patients with prior injuries to study knee
* Patients with history of childhood knee disease
* Patients who cannot complete questionnaires in English
* Patients with comorbidities preventing surgery
* Patients who are not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Jr Score | Baseline, 2 weeks post op, 6 weeks post op, 1 week post op
  The KOOS Jr Score is a patient-reported outcome measure, scaled from 0-28, with higher scores meaning worse outcomes.

SECONDARY OUTCOMES:
Patient Reported Outcome Measure Information System (PROMIS) Physical Function | Baseline, 2 weeks post op, 6 weeks post op, 1 week post op
  The PROMIS Physical Function Score is a patient-reported outcome measure, scaled from 0-20, with higher scores meaning improved outcomes.

OTHER OUTCOMES:
Patient Reported Outcome Measure Information System (PROMIS) Pain Interference | Baseline, 2 weeks post op, 6 weeks post op, 1 week post op
  The PROMIS Pain Interference Score is a patient-reported outcome measure, scaled from 0-20, with higher scores meaning worse pain.
Forgotten Joint Score | Baseline, 2 weeks post op, 6 weeks post op, 1 week post op
  The Forgotten Joint Score is a patient-reported outcome measure, scaled from 0-100, with higher scores meaning improved outcomes.
Pain Visual Analogue Scale | Baseline, 2 weeks post op, 6 weeks post op, 1 week post op
  Pain scale scaled from 0-10 with higher scores indicating more pain.
Range of motion | Baseline, 2 weeks post op, 6 weeks post op, 1 week post op
  Range of motion defined as degrees of knee extension and flexion

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Brown, MD, Principal Investigator — Loyola University Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blakeney W, Clement J, Desmeules F, Hagemeister N, Riviere C, Vendittoli PA. Kinematic alignment in total knee arthroplasty better reproduces normal gait than mechanical alignment. Knee Surg Sports Traumatol Arthrosc. 2019 May;27(5):1410-1417. doi: 10.1007/s00167-018-5174-1. Epub 2018 Oct 1. PMID 30276435
- [Background] Elbuluk AM, Jerabek SA, Suhardi VJ, Sculco PK, Ast MP, Vigdorchik JM. Head-to-Head Comparison of Kinematic Alignment Versus Mechanical Alignment for Total Knee Arthroplasty. J Arthroplasty. 2022 Aug;37(8S):S849-S851. doi: 10.1016/j.arth.2022.01.052. Epub 2022 Jan 31. PMID 35093548
- [Background] Jaffe WL, Dundon JM, Camus T. Alignment and Balance Methods in Total Knee Arthroplasty. J Am Acad Orthop Surg. 2018 Oct 15;26(20):709-716. doi: 10.5435/JAAOS-D-16-00428. PMID 30134305
- [Background] Lee YS, Howell SM, Won YY, Lee OS, Lee SH, Vahedi H, Teo SH. Kinematic alignment is a possible alternative to mechanical alignment in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3467-3479. doi: 10.1007/s00167-017-4558-y. Epub 2017 Apr 24. PMID 28439636
- [Background] Li Y, Wang S, Wang Y, Yang M. Does Kinematic Alignment Improve Short-Term Functional Outcomes after Total Knee Arthroplasty Compared with Mechanical Alignment? A Systematic Review and Meta-analysis. J Knee Surg. 2018 Jan;31(1):78-86. doi: 10.1055/s-0037-1602136. Epub 2017 May 1. PMID 28460408
- [Background] Luceri F, Sosio C, Sirtori P, Battistella D, Zuffada M, Ulivi M, Meroni V, Marmotti A, Mangiavini L, Peretti GM. Kinematic versus mechanical alignment in total knee arthroplasty: a preliminary study. J Biol Regul Homeost Agents. 2020 Jul-Aug;34(4 Suppl. 3):139-143. Congress of the Italian Orthopaedic Research Society. PMID 33261269
- [Background] Luo Z, Zhou K, Peng L, Shang Q, Pei F, Zhou Z. Similar results with kinematic and mechanical alignment applied in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2020 Jun;28(6):1720-1735. doi: 10.1007/s00167-019-05584-2. Epub 2019 Jun 27. PMID 31250055
- [Background] McEwen PJ, Dlaska CE, Jovanovic IA, Doma K, Brandon BJ. Computer-Assisted Kinematic and Mechanical Axis Total Knee Arthroplasty: A Prospective Randomized Controlled Trial of Bilateral Simultaneous Surgery. J Arthroplasty. 2020 Feb;35(2):443-450. doi: 10.1016/j.arth.2019.08.064. Epub 2019 Sep 5. PMID 31591010
- [Background] Oussedik S, Abdel MP, Victor J, Pagnano MW, Haddad FS. Alignment in total knee arthroplasty. Bone Joint J. 2020 Mar;102-B(3):276-279. doi: 10.1302/0301-620X.102B3.BJJ-2019-1729. PMID 32114811
- [Background] Riviere C, Iranpour F, Auvinet E, Howell S, Vendittoli PA, Cobb J, Parratte S. Alignment options for total knee arthroplasty: A systematic review. Orthop Traumatol Surg Res. 2017 Nov;103(7):1047-1056. doi: 10.1016/j.otsr.2017.07.010. Epub 2017 Aug 31. PMID 28864235
- [Background] Tian G, Wang L, Liu L, Zhang Y, Zuo L, Li J. Kinematic alignment versus mechanical alignment in total knee arthroplasty: An up-to-date meta-analysis. J Orthop Surg (Hong Kong). 2022 Sep-Dec;30(3):10225536221125952. doi: 10.1177/10225536221125952. PMID 36250421
- [Background] Weber P, Gollwitzer H. Kinematic alignment in total knee arthroplasty. Oper Orthop Traumatol. 2021 Dec;33(6):525-537. doi: 10.1007/s00064-021-00729-4. Epub 2021 Aug 19. PMID 34414467